CLINICAL TRIAL: NCT05095675
Title: Predicting Effective Adaptation to Breast Cancer to Help Women to BOUNCE Back: a Multicentre Clinical Pilot Study
Brief Title: Predicting Effective Adaptation to Breast Cancer to Help Women to BOUNCE Back
Acronym: BOUNCE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: European Institute of Oncology (Other)
Collaborators: Helsinki University Central Hospital (Other); Hebrew University of Jerusalem (Other); Fundacao Champalimaud (Other); Foundation for Research and Technology - Hellas (Unknown); Institute of Communications and Computer Systems, Athens, Greece (Other); SINGULARLOGIC (Unknown); NHG CONSULTING OY (Unknown); Noona Healthcare (Unknown)
Responsible Party: Sponsor
Other Study IDs: R868/18-IEO 916
Record Dates: First submitted 2021-01-20; First posted 2021-10-27 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
Keywords: Resilience; Predictive model
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: psychological questionnaires — Participants have to fulfill psychological questionnaires in different time points during medical oncological treatment

SUMMARY:
Breast cancer accounts for 28% of all cancer cases in Europe ("WHO," 2018). Coping with breast cancer is becoming an increasingly burdensome socio-economic challenge, partly due to the increasing incidence registered in the last years, which is occurring despite continuous advances in medicine. This said, mortality rate has decreased significantly as 5-year survival rate has risen from 75% to 90% ("Breast Cancer Research Foundation," 2016). For these reasons the number of cancer survivors has grown, with important effects on quality of life even years after the end of treatments.

The process of successful adaptation to breast cancer and the various accompanying stressors can be conceptually defined as the person's resilience. Resilience is a complex construct that can be defined on different levels: an individual's potential (capacity to engage in adaptive coping processes), a process (adaptive reactions to adversity), and an outcome (the final state achieved as the result of coping).

While theoretical contributions regarding resilience models in medical settings have been advanced (Deshields et al., 2016), to date no one has tested the integrated contributing role of multiple psychological, biological and functional variables in predicting the patient's ability to bounce back from the stressful life event of being diagnosed with breast cancer. Resilience is going to be measured through a data-driven method (computation of resilience index on the basis of retrospective data) and through a psychometric method (various domains of resilience through questionnaires).

There is a growing need for novel strategies to improve the understanding and the capacity to predict resilience of women to the variety of stressful experiences.

BOUNCE European Project (H2020 European Project "Predicting Effective Adaptation to Breast Cancer to Help Women to BOUNCE back"; Grant Agreement Nr: 777167) will bring together modelling, medical, and social sciences experts to advance current knowledge on the dynamic nature of resilience as it relates to improved quality of life.

The broad and general objective of the BOUNCE project is to build a quantitative mathematical model of factors associated with optimal adjustment capacity to cancer. The investigators will collect biomedical status (BMS), the psychosocial status (PSS) and the functional status (FUS) of breast cancer patients that literature demonstrated to be predictive of patients' capacity to bounce back during the highly stressful treatment and recovery period following diagnosis of breast cancer. The overarching goal of the model is to understand which factors predict optimal adjustment to breast cancer and which combination of factors undermine adjustment. This would allow early identification of women at risk for which it is better to intervene through a personalised psychological support.

Funding: The BOUNCE Project "Predicting Effective Adaptation to Breast Cancer to Help Women to BOUNCE back" has received funding from the European Union's Horizon 2020 research and innovation programme, Project type: H2020 - SCI-2017-CNECT-2; Project type: H2020 - SCI-2017-CNECT-2; Grant Agreement Nr: 777167.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a devoted informed consent signed by the patient and the physician
* Histologically confirmed invasive early or locally advanced operable breast cancer
* Tumour stage I, II and III
* Patients receiving surgery as part of the local treatment
* Patients receiving any type of systemic treatment regardless of treatment type and/or adjuvant radiation therapy if indicated as part of the local treatment

Exclusion Criteria:

* Refusal to sign informed consent
* Presence of distant metastases
* History of another malignancy or contralateral invasive breast cancer within the last five years except cured basal cell carcinoma of skin or carcinoma in situ of the uterine cervix
* History of early onset (i.e., before 40 years of age) mental disorder (i.e., schizophrenia, psychosis, bipolar disorder, diagnosis of major depression) or severe neurologic disorder (i.e., neurodegenerative disorder, dementia)
* Serious other diagnosed concomitant diseases such as clinically significant (i.e. active) cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease or cardiac arrhythmia not well controlled with medication) or myocardial infarction within the last 12 months.
* Major surgery for a severe disease or trauma which could affect patient's psychosocial wellbeing (for example, major heart or abdominal surgery) within 4 weeks prior to study entry or lack of complete recovery from the effects of surgery
* Treatment for invasive cancer
* Treatment for any major illness in the last half year
* Pregnancy or breastfeeding at time of recruitment

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are breast cancer patients with stage I-III histologically confirmed diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 660 (Estimated)
Dates: Start 2018-12-06 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Resilience | Every 3 months, until completion of the study, on average 2 years
  Assessed by the Connor Davidson Resilience Scale (CD-RISC). The scale consists in ten item on a 5-point Likert scale, ranging from 0 (not true at all) to 4 (true nearly all the time).
Personality | one measurement at Day 1
  Assessed by the Ten Item Personality Inventory (TIPI). The scale consists in 10-item (measure of the Big Five dimensions) on a 7-point Likert scale, ranging from 1(Disagree strongly) to 7 (Agree strongly)
Dispositional optimism | one measurement at Day 1
  Assessed by the Life Orientation Test-Revised (LOT-R). The scale is a 10-item scale that measures optimistic and pessimistic disposition. Respondents use a 5-point rating scale (0 = strongly disagree; 4 = strongly agree) to show how much they agree with 10 statements about positive and negative expectations.
Sense of coherence | one measurement at Day 1
  Assessed by the Sense of Coherence (SOC) 13 item scale. The response alternatives are a semantic scale of 1 point to 7 points, where 1 and 7 indicate extreme feelings about questions (and statements) about how one's life is experienced
Change in Post traumatic stress disorder | Every 3 months, until completion of the study, on average 2 years
  Assessed by the PCL-5. The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. Respondents use a 5-point Likert scale (0 = "Not at all" to 4 = "Extremely")
Change in Positive outcome after trauma exposure | Every 3 months, until completion of the study, on average 2 years
  Assessed by the Posttraumatic Growth Inventory (PTGI)10 item, developed to assess growth following traumatic events. The scale consists on a 6-point Likert scale
Change in Coping flexibility | Every 3 months, until completion of the study, on average 2 years
  Assessed by the Perceived ability to cope with trauma (PACT). The questionnaire has two scales that measure the perceived ability to focus on processing the trauma (trauma focus) and to focus on moving beyond the trauma (forward focus). Respondents use a 7-point scale ranging from 1 (not at all able) to 7 (extremely able)
Change in Cognitive coping strategies | Every 3 months, until completion of the study, on average 2 years
  Assessed by the Cognitive Emotion Regulation Questionnaire 18 items(CERQ). The questionnaire is constructed in order to identify the cognitive emotion regulation strategies used after a negative events or situations. Responsens are given on a 5-point Likert scale ranging from 1 (almost never) to 5 (almost always).
Change in Dispositional mindfulness | Every 3 months, until completion of the study, on average 2 years
  Assessed by the Mindful attention awareness scale (MAAS). The scale consists in 15 item (1-6 Likert scale, from 1 "almost always" to 6 "almost never" ) designed to assess open or receptive awareness of and attention to what is taking place in the present.
Change in Mental adjustment to cancer | Every 3 months, until completion of the study, on average 2 years
  Assessed by the mini mental adjustment to cancer (mini-MAC). The scale consists in 29 statements allowing the identification and evaluation of four types of strategies of coping with disease. The mini-MAC scale is a self-descriptive tool. The respondent use a four-point scale, to what extent a given statement applies at present.
Change in Social support | Every 3 months, until completion of the study, on average 2 years
  Assessed by the modified Medical Outcome Study -Social Support survey(mMOS-SS). The mMOS-SS assess the emotional and the instrumental social support.
  The Mini-MAC items are rated on a 4-point Likert scale ranging from "Definitely does not apply to me" (1) to "Definitely apply to me" (4).
Change in Family resilience | Every 3 months, until completion of the study, on average 2 years
  Assessed by the Family resilience questionnaire (F.A.R.E). The FaRE Questionnaire is designed to measure family resilience in oncological settings. The scale has 24 item on a 7-point Likert scale (from strongly agree to strongly disagree).
Change in Illness representation | Every 3 months, until completion of the study, on average 2 years
  Assessed by the Illness perception questionnaire revised (IPQ-r). The illness perceptions questionnaire measures an individual's beliefs and feelings about their illness. The scale consists in 84 items on a 5-point Likert style scale, ranging from strongly disagree to strongly agree.
Change in patients Self-efficacy in coping with cancer | Every 3 months, until completion of the study, on average 2 years
  Assessed by the Cancer behavior inventory-brief (CBI-B), a measure of self-efficacy for coping in cancer patients. The instrument consists of 12 items (rated 1 = not at all confident to 7 = totally confident).
Change in Depression and anxiety | Every 3 months, until completion of the study, on average 2 years
  Assessed by the Hospital Anxiety and Depression Scale (HADS). is a 14-item self-report measure designed to assess depression and anxiety. Respondents are asked to rate each statement in considering the previous week on a 0-4 scale that taps into frequency.
Change in Quality of life assessed by EORTC-QLQ C30 | Every 3 months, until completion of the study, on average 2 years
  Assessed by the European Organization for Research and Treatment of Cancer quality of life questionnaire-Core 30 (EORTC QLQ-C30). The EORTC QLQ-C30 includes 30 items that are rated on a 4-point scale that ranges from 1 "not at all" to 4 "very much". The EORTC QLQ-C30 has a global score, 5 functional scales (physical, role, emotional, cognitive and social), 3 symptoms scales (fatigue, nausea/vomiting, pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties).
Change in Quality of life in patients with breast cancer assessed by EORTC-QLQ BR23 | Every 3 months, until completion of the study, on average 2 years
  Assessed by the European Organization for Research and Treatment of Cancer (EORTC) Breast Cancer-Specific Quality of Life Questionnaire (QLQ-BR23. The scale consists in 23 item on a likert scale from 1 "not at all" to 4 "very much", assessing body image, sexual functioning, sexual enjoyment, future perspective, systemic therapy side effects, breast symptoms, arm symptoms and upset by hair loss.
Change in Fear of cancer recurrence | Every 3 months, until completion of the study, on average 2 years
  Assessed by the Fear of Cancer Recurrence Inventory-Short Form (FCRI-SF). The scale consists in 9 items rated on a Likert scale ranging from 0 ("not at all" or "never") to 4 ("a great deal' or "all the time").
Change in Positive and negative affect | Every 3 months, until completion of the study, on average 2 years
  Assessed by the Positive and Negative Affect Schedule-short form (PANAS-FS). The scale consists of two 5-item scales to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much).
Change in Distress | Every 3 months, until completion of the study, on average 2 years
  Assessed by the Distress Thermometer (DT). The scale consists in a single-item tool using a 0 (no distress) to 10 (extreme distress)-point Likert scale resembling a thermometer. The patient rates the level of distress over the past week.

SECONDARY OUTCOMES:
Chronic illnesses | one measurement at Day 1
  assessed by the presence of comorbidity (yes/no)
Genetic risk factors | one measurement at Day 1
  assessed by the presence of family history of first-degree relative's breast cancer and presence of mutation (yes/no)
Change in Menopausal status | at Day 1 and after one year
  assessed by one of the following categories: Premenopausal Perimenopausal Postmenopausal
Tumor biology | one measurement at Day 1
  assessed by indicating the following clinical characteristics: pT (mm) pN (N1,N2,N3) Histological type (ductal, lobular, other) ER (%) PR (%) Grade (I, II,III) HER2 positive or negative (FISH, SISH/CISH)
surgery type | after six months
  assessed using one of the following categories: quadrantectomy or mastectomy, axillary dissection or sentinel lymph node biopsy
Change in Performance status | every 3 month until one year
  assessed by using the ECOG scale
Change in Ongoing oncological therapy | every 6 month until completion of the study, on average 2 years
  assessed by indicating the type of oncological treatment using one of the following categories: chemotherapy, radiotherapy, endocrine therapy or Anti HER2 therapy
Change in the use of Psychotropic medication | every 3 month until completion of the study, on average 2 years
  assessed by indicating the type of the Psychotropic medication prescribed to the patient
Change in blood test | at Day 1 and after 12 months
  assessed by the following Laboratory tests: hemoglobin (gdl), leukocytes (10*3 mcl), thrombocytes (10*3 mcl), neutrophils (%), hs-CRP(number)
Age | one measurement at Day 1
  assessed in years
Change in Level of education | At Day 1 and at up to 2 years
  Assessed by the highest level of education indicated by patients using one of the following categories: Primary school, Secondary school, High school, Vocational non-academic diploma, Bachelor degree, Postgraduate education (Master degree, PhD, Nba, specialization, etc.,)
Change in Marital status | At Day 1 and up to 2 years
  assessed by the type of civil status indicated by patients using one of the following categories: Single, Engaged, Common-law partner, Married, Separated/divorced, Widowed
Change in Weight | Every 6 months, until completion of the study, on average 2 years
  assessed by kilograms
Change in Height | Every 6 months, until completion of the study, on average 2 years
  assessed by centimeters
Change in Number of children | At Day 1 and up to 2 years
  assessed by the number of children declared by patients
Change in Employment status | Every 3 months, until completion of the study, on average 2 years
  assessed by occupational status indicating by patients using one of the following categories: Employed full time, Employed part time, Self-employed, Unemployed, Retired, Housewife
Change in number of sick days | Every 3 months, until completion of the study, on average 2 years
  assessed by the number of workdays missed because of illness or treatments declared by patients
Change in Flexible arrangements at work | After one year and up to 2 years
  assessed by asking patients if they had support from employer to obtain more flexible work arrangements
Return to work | up to 2 years
  assessed by asking patients if they returned to work
Change in monthly Income | At Day 1 and up to 2 years
  assessed by asking patients to indicate monthly income using one of the following categories: 0-500; 501-1,000; 1,001-1,500; 1,501-2,000; 2,001-2,500; 2,501-3,000; 3,001-3,500; 3,501-4,000; 4,001-4,500; 4,501 and up
Change in level of faith | At Day 1 and up to 2 years
  assessed by asking patients to describe religion faith using the following categories: Ateist, Practicing believer, Non-practicing believer,
Change in Number of professional support sessions | Every 3 months, until completion of the study, on average 2 years
  assessed by asking patients if they met mental health professional
Change in family's work | Every 3 months, until completion of the study, on average 2 years
  assessed by asking patients if their partner or someone in their family reduced their work time to take care of the patient
Change in leisure activities | Every 3 months, until completion of the study, on average 2 years
  assessed by asking patients to indicate if they are engaged in some activities to support well-being (e.g. culture&arts, other hobbies, mindfulness/yoga, etc)
Change in domestic help | Every 3 months, until completion of the study, on average 2 years
  assessed by number of days declared by patients
Change in Smoking habits | At Day 1, after 9 months and up to 2 years
  assessed by the number of smoked cigarettes
Change in alcohol consumption | At Day 1, after 9 months and up to 2 years
  assessed by asking patients how often they drink alcohol using one of the following categories: Never, Less than once a month, Once or twice a month, About once a week, Several times a week, Every day
Change in Drug use | Every 6 months, until completion of the study, on average 2 years
  assessed by asking patients if they use drugs and the type of drugs using one of the following categories: No, Not medically-prescribed drugs (such as tranquilizers, Ritalin or strong pain-killers), Medically-prescribed cannabis, Not medically-prescribed cannabis, Other drugs (such as MDMA or cocaine)
Change in diet habits | At Day 1, after 9 months and up to 2 years
  assessed by asking patients if they followed a specific diet and what type of diet, using one of the following categories: Low-calories, Low-carb, Mediterranean, Protein-only, Vegan, Vegeterian, Gluten-free, Dairy-free, FODMAP-free, Macrobiotic diet, Other, please specify
Change in Physical exercise | Every 6 months, until completion of the study, on average 2 years
  assessed by asking patients the type and the amount of physical excercise using one of the following categories: Moderate aerobic exercise (for example walking, cycling) in min/week; Heavy aerobic exercise (for example running, HIIT training) in min/week; Muscle training in times/week; no exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Ketti Mazzocco, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy

REFERENCES:
- [Derived] Karademas EC, Roziner I, Mazzocco K, Pat-Horenczyk R, Sousa B, Oliveira-Maia AJ, Stamatakos G, Kondylakis H, Kolokotroni E, Almeida S, Lemos R, Mattson J, Simos P, Poikonen-Saksela P. The illness representations-physical well-being interplay over time in breast cancer patients. Health Psychol. 2025 Aug;44(8):779-788. doi: 10.1037/hea0001499. Epub 2025 Mar 27. PMID 40146609
- [Derived] Dahabre R, Bentley G, Poikonen-Saksela P, Mazzocco K, Sousa B, Pat-Horenczyk R. Can mindfulness facilitate posttraumatic growth in breast cancer patients? The mediating role of illness perceptions and positive emotions. J Health Psychol. 2024 Apr;29(5):438-451. doi: 10.1177/13591053231223484. Epub 2024 Feb 5. PMID 38312012
- [Derived] Pettini G, Sanchini V, Pat-Horenczyk R, Sousa B, Masiero M, Marzorati C, Galimberti VE, Munzone E, Mattson J, Vehmanen L, Utriainen M, Roziner I, Lemos R, Frasquilho D, Cardoso F, Oliveira-Maia AJ, Kolokotroni E, Stamatakos G, Leskela RL, Haavisto I, Salonen J, Richter R, Karademas E, Poikonen-Saksela P, Mazzocco K. Predicting Effective Adaptation to Breast Cancer to Help Women BOUNCE Back: Protocol for a Multicenter Clinical Pilot Study. JMIR Res Protoc. 2022 Oct 12;11(10):e34564. doi: 10.2196/34564. PMID 36222801